CLINICAL TRIAL: NCT05949190
Title: Improving Cognition and Gestational Duration With Targeted Nutrition
Acronym: COGENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Open Philanthropy (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); Ministry of Health and Sanitation, Sierra Leone (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 202305139
Record Dates: First submitted 2023-06-29; First posted 2023-07-17 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition in Pregnancy; Preterm Birth; Child Development; Postpartum Depression; Antepartum Depression
MeSH Terms: conditions — Premature Birth; Depression, Postpartum | interventions — Azithromycin; Albendazole; fanasil, pyrimethamine drug combination; Cognitive Behavioral Therapy; Insecticide-Treated Bednets

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In the food comparison, while the 2 study foods taste similar, full masking cannot be guaranteed. In the CBT comparison, participants and therapists will not be masked. In all cases, outcomes assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) and CBT (Experimental): Factorial 1. A daily dose of 500mg DHA, 500mg EPA, and 550mg choline will be added to the maternal balanced energy-protein RUSF. One sachet (daily dose) will provide 520 Kcal, 18g protein, and the same quantities of micronutrients as the United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) for women. M-RUSF+ will be vacuum sealed and packaged in foil sachets containing 100g of food.
  Factorial 2. Among participants randomized to receive M-RUSF+ vs. M-RUSF, those who develop ante- or postpartum depression will receive 6 sessions of CBT adopted for use in illiterate populations will be provided.
  Interventions: Dietary Supplement: M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline); Drug: Azithromycin; Drug: Albendazole; Drug: Sulfadoxine pyrimethamine; Behavioral: Cognitive behavioral therapy; Other: Insecticide-treated mosquito net
- M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) and no CBT (Experimental): Factorial 1. A daily dose of 500mg DHA, 500mg EPA, and 550mg choline will be added to the maternal balanced energy-protein RUSF. One sachet (daily dose) will provide 520 Kcal, 18g protein, and the same quantities of micronutrients as the UNICEF/World Health Organization/United Nations multiple micronutrient supplement for pregnant/lactating women. M-RUSF+ will be vacuum sealed and packaged in foil sachets containing 100g of food.
  Factorial 2. Participants who develop ante- or postpartum depression will not receive CBT.
  Interventions: Dietary Supplement: M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline); Drug: Azithromycin; Drug: Albendazole; Drug: Sulfadoxine pyrimethamine; Other: Insecticide-treated mosquito net
- M-RUSF (Maternal Ready-to-use Supplementary Food without DHA/EPA/choline and CBT (Experimental): Factorial 1. M-RUSF will be similar to M-RUSF+, except it will not contain added DHA or EPA, and will only contain 5mg of added choline to help with flavor masking. One sachet (daily dose) will provide 520 Kcal, 18g protein, and the same quantities of micronutrients as the UNIMMAP for pregnant/lactating women. M-RUSF+ will be vacuum sealed and packaged in foil sachets containing 100g of food.
  Factorial 2. Participants who develop ante- or postpartum depression will receive 6 sessions of CBT adopted for use in illiterate populations will be provided.
  Interventions: Dietary Supplement: M-RUSF (Maternal Ready-to-Use Supplementary Food); Drug: Azithromycin; Drug: Albendazole; Drug: Sulfadoxine pyrimethamine; Behavioral: Cognitive behavioral therapy; Other: Insecticide-treated mosquito net
- M-RUSF (Maternal Ready-to-use Supplementary Food without DHA/EPA/choline and no CBT (Experimental): Factorial 1. M-RUSF will be similar to M-RUSF+, except it will not contain added DHA or EPA, and will only contain 5mg of added choline to help with flavor masking. One sachet (daily dose) will provide 520 Kcal, 18g protein, and the same quantities of micronutrients as the UNIMMAP for pregnant/lactating women. M-RUSF+ will be vacuum sealed and packaged in foil sachets containing 100g of food.
  Factorial 2. Participants who develop ante- or postpartum depression will not receive CBT.
  Interventions: Dietary Supplement: M-RUSF (Maternal Ready-to-Use Supplementary Food); Drug: Azithromycin; Drug: Albendazole; Drug: Sulfadoxine pyrimethamine; Other: Insecticide-treated mosquito net

INTERVENTIONS:
Dietary Supplement: M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) — Balanced energy protein supplement with added DHA/EPA/choline, micronutrients
  Arms: M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) and CBT; M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) and no CBT
Dietary Supplement: M-RUSF (Maternal Ready-to-Use Supplementary Food) — Balanced energy protein supplement with added micronutrients
  Arms: M-RUSF (Maternal Ready-to-use Supplementary Food without DHA/EPA/choline and CBT; M-RUSF (Maternal Ready-to-use Supplementary Food without DHA/EPA/choline and no CBT
Drug: Azithromycin — 1g dose
Drug: Albendazole — 400mg dose
Drug: Sulfadoxine pyrimethamine — Monthly, 1,500/75mg dose
Behavioral: Cognitive behavioral therapy — Novel program developed for illiterate end-users
  Arms: M-RUSF (Maternal Ready-to-use Supplementary Food without DHA/EPA/choline and CBT; M-RUSF+ (Maternal Ready-to-Use Supplementary Food + DHA/EPA/choline) and CBT
Other: Insecticide-treated mosquito net — Bed net to prevent malaria

SUMMARY:
The goal of this clinical trial is to test (1) a novel maternal ready-to-use supplementary food and (2) a novel cognitive behavioral therapy intervention in undernourished Sierra Leonean women. The main questions it aims to answer are:

* Will the addition of omega-3 long-chain polyunsaturated fatty acids docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), as well as choline, to a maternal ready-to-use supplementary food (M-RUSF+) prolong gestation when compared with a similar supplementary food except that it lacks DHA, EPA, and choline (M-RUSF)?
* Will M-RUSF+ improve infant cognitive development at 9 months of age when compared with M-RUSF?
* Will the novel CBT program improve ante- and post-partum depression?

DETAILED DESCRIPTION:
Undernutrition in pregnancy is common, affecting nearly 10% of women worldwide and 25% of women in Sub-Saharan Africa, and increases risks for both mothers and their offspring, including bleeding, preterm birth, neonatal mortality, and impaired infant cognitive development. Available treatments have limited impact on these outcomes, which affect millions annually. A recent trial in Sierra Leone showed that pairing high-quality supplementary nutrition with anti-infective measures led to greater maternal weight gain, longer and heavier newborns, and reduced neonatal mortality. In addition, ante- and postpartum depression are underrecognized and undertreated in rural Sub-Saharan Africa.

The goal of this clinical trial is to test (1) a novel maternal ready-to-use supplementary food (M-RUSF+) and (2) a novel cognitive behavioral therapy (CBT) program developed for illiterate users, in undernourished pregnant women in Sierra Leone. The main questions it aims to answer are:

* Will the addition of omega-3 long-chain polyunsaturated fatty acids docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), as well as choline, to a maternal ready-to-use supplementary food (M-RUSF+) prolong gestation when compared with a similar supplementary food except that it lacks DHA, EPA, and choline (M-RUSF)?
* Will M-RUSF+ improve infant cognitive development at 9 months of age when compared with M-RUSF?
* Will the novel CBT program improve ante- and post-partum depression?

Participants will present to government-run antenatal clinics for screening. If they quality for enrollment and consent to participate, they will undergo:

ANTENATALLY

* randomization to intervention vs. control group
* bi-weekly anthropometric measurements
* ultrasound gestational age estimation
* demographic, socioeconomic, and health history questionnaires
* bi-weekly blood pressure measurement
* bi-weekly screening for ante- and post-partum depression
* two blood spot collections

POSTNATALLY

* birth measurements of mother and offspring
* cord blood and placental sampling for a subset
* 5 clinic visits for mother and offspring anthropometric measurements, health history, breastfeeding practice, maternal mental health questions
* offspring developmental assessments

All participants will receive:

ANTENATALLY

* 100g/day of M-RUSF+ or M-RUSF, containing 530 Kcal, 19g protein, United Nations International Multiple Micronutrient Antenatal Preparation (UNIMMAP) equivalent
* insecticide-treated bed nets
* a single dose of albendazole de-worming medicine
* monthly malaria chemoprophylaxis
* single doses of azithromycin in the second and third trimesters
* safe birth kits

If participants develop ante- or postpartum depression and are randomized to CBT, they will receive 6 sessions of CBT.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the M-RUSF+ vs. M-RUSF element of the study, an individual must meet all of the following criteria:

1. Provision of signed (or thumb-printed) and dated informed consent form 1a. Women who are ≥ 18 years of age or married will be allowed to consent for themselves 1b. Women who are < 18 years of age and unmarried must provide assent and a parent or guardian must provide consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study, including no plan to move from the catchment area of a participating clinic
3. ≥ 13 years of age
4. Pregnant
5. Mid-upper arm circumference ≤ 23 cm or body-mass index < 18.5

In order to be eligible to participate in the CBT vs. no CBT element of the study (factorial design with the above), an individual must be enrolled in the M-RUSF+ vs. M-RUSF study and meet the following criteria:

1. Provision of signed (or thumb-printed) and dated informed consent form 1a. Women who are ≥ 18 years of age or married will be allowed to consent for themselves 1b. Women who are < 18 years of age and unmarried must assent and a parent or guardian consent must provide consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study, including no plan to move from the catchment area of a participating clinic
3. Patient Health Questionnaire-9 score ≥ 9

Exclusion Criteria:

1. Participation in a concomitant supplementary feeding program
2. Known allergy to components of intervention or control study food or medications
3. Known gestational diabetes
4. Hypertension
5. Severe anemia, or other condition requiring immediate hospitalization

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Gestational duration | Enrollment to birth (range 2 to 26 weeks)
  Enrollment ultrasound estimated gestational age plus time between enrollment and delivery. For the primary outcome, this will only be assessed among participants enrolled <= 30 weeks gestational age and with singleton live births
Malawi Developmental Assessment Tool (MDAT) global z-score | 9 months post-birth
  Infant global age-adjusted z-score on MDAT
Adapted Patient Health Questionnaire-9 (PHQ-9) score | 8 weeks after diagnosis with ante- or post-partum depression
  Among participants who develop ante- or post-partum depression, adapted Patient Health Questionnaire-9 score, (range 0-27, higher scores are worse)

SECONDARY OUTCOMES:
Early preterm birth | Enrollment to 34 weeks' gestation
  Birth < 34 weeks gestational age
Birth weight | Birth
  Infant weight at birth
Birth length | Birth
  Infant length at birth
Low birth weight | Birth
  Birth weight < 2.5 kg
Malawi Developmental Assessment Test sub-domain z-scores | 9 months after birth
  Gross motor, fine motor, language, and social domain z-scores (expected range -4 to 2, higher scores are better)
Preterm birth | Enrollment to 37 weeks' gestation
  Birth < 37 weeks gestational age
Neonatal mortality | Birth to 28 days of age
  Infant death within the first 28 days of life
Infant mortality | Birth to end of follow-up (9 months)
  Infant death
Depressive symptoms | Through study completion, an average of 1.25 years
  Adapted Patient Health Questionnaire-9 score (range 0-27, higher scores are worse)
Maternal and infant DHA status | From Enrollment to delivery, an average of 15 weeks
  Maternal plasma, cord blood DHA status
Maternal and infant choline status | From Enrollment to delivery, an average of 15 weeks
  Blood choline concentration
Maternal weight gain | From Enrollment to delivery, an average of 15 weeks
  Average weekly weight gain
Post-term delivery | From Enrollment to delivery, an average of 15 weeks
  Delivery > 42 weeks' gestation
Depression incidence | 8 weeks from time of depression diagnosis
  Adapted PHQ-9 >= 9
Birth chest circumference | Birth
  Infant chest circumference
Birth thigh circumference | Birth
  Infant thigh circumference
Birth head circumference | Birth
  Infant head circumference
Infant weight at 6 weeks, 3 months, 6 months, 9 months | Birth to 9 months
  Infant weight
Infant length at 6 weeks, 3 months, 6 months, 9 months | Birth to 9 months
  Infant length
Infant length-for-age z-score at 6 weeks, 3 months, 6 months, 9 months | Birth to 9 months
  Infant length-for-age z-score
Gestational duration | From Enrollment to birth, an average of 15 weeks
  Enrollment ultrasound estimated gestational age plus time between enrollment and delivery. For this secondary outcome, all enrolled women will be included in analysis.
Placental weight | Birth
  Weight of placenta in grams
Small for gestational age (SGA) | Birth
  Under 10th percentile in birth weight for gestational age

OTHER OUTCOMES:
Intrauterine growth parameters | Subset of participants (enrollment GA <= 24 weeks) to undergo q4-6week serial ultrasounds
  Estimated weight, head circumference, femur length, placental size
Gestational duration by baseline DHA status | From enrollment to birth, an average of 15 weeks
  Gestational duration modeled by enrollment DHA % of plasma fatty acids
Gestational duration by baseline maternal MUAC | From enrollment to birth, an average of 15 weeks
  Gestational duration modeled by enrollment MUAC
Gestational duration by enrollment gestational age | From enrollment to birth, an average of 15 weeks
  Gestational duration modeled by enrollment GA
Gestational duration by enrollment maternal age | From enrollment to birth, an average of 15 weeks
  Gestational duration modeled by enrollment maternal age
Gestational duration by maternal parity | From enrollment to birth, an average of 15 weeks
  Gestational duration compared across levels of maternal parity

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- Sierra Leone (10):
  - Bandajuma, Bandajuma, Southern Province
  - Bendu Malen, Bendu, Southern Province
  - Blama Massaquoi, Blama Massaquoi, Southern Province
  - Futa Peje, Futa Peje, Southern Province
  - Gbondapi, Gbondapi, Southern Province
  - Nyandehun Malen, Nyandehun, Southern Province
  - Potoru, Potoru, Southern Province
  - Pujehun Static, Pujehun, Southern Province
  - Sahn Malen, Sahn, Southern Province
  - Zimmi, Zimmi, Southern Province

IPD SHARING:
Plan to Share IPD: Yes
All collected Individual; Patient Data (IPD).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 12 months of primary publication